CLINICAL TRIAL: NCT01854580
Title: Evaluation of an Integrated Care Project of the Statutory Health Insurance Techniker Krankenkasse [Evaluation Des Integrierten Versorgungsangebots Der Techniker Krankenkasse]
Brief Title: Evaluation of an Integrated Care Project
Acronym: ediva
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med, MBA, Charite University, Berlin, Germany
Other Study IDs: 1-Witt
Record Dates: First submitted 2013-04-22; First posted 2013-05-15 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Asthma; Allergic Rhinitis; Atopic Eczema; Migraine; Headache; Depression
Keywords: Comparative effectiveness research; health economic evaluation
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Dermatitis, Atopic; Migraine Disorders; Headache; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Integrated care: Insured people in the Techniker Krankenkasse that are registered in the integrated care project.
- Control group: Insured people in the Techniker Krankenkasse that are not registered in the integrated care project.

SUMMARY:
The purpose of the study is to investigate the effectiveness and cost-effectiveness of the integrated care program of a statutory health insurance offering additional homeopathic treatment to their members

DETAILED DESCRIPTION:
The German statutory health insurance 'Techniker Krankenkasse' offers an integrated additional homeopathic treatment. To date, this offer has not been evaluated. Therefore we aim to investigate the effectiveness as well as the cost-effectiveness of this program in adolescents (12-17 years) and adults with various chronic diseases.

In an observational study we plan to compare patients participating in the integrated care project with matched insured persons from the Techniker Krankenkasse that do not participate in this program.

Matching will be based on gender, age and diagnosis. Regarding the diagnosis, we plan to include adolescents with: asthma, allergic rhinitis and atopic eczema; and adults with asthma, allergic rhinitis and atopic migraine, headache and depression.

To measure effectiveness, patients have to complete diagnosis-specific questionnaires at baseline and 3, 6 and 12 months. The primary outcome for each diagnosis is measured with diagnosis-specific questionnaire at 6 months. Secondary outcomes include quality of life (SF-12) at 3, 6 and 12 months as well as the diagnosis-specific questionnaires at 3 and 12 months.

ELIGIBILITY:
Inclusion criteria:

* Newly registered for the integrated care program
* Insured for at least 1 year at the Techniker Krankenkasse
* Having access to the internet and e-mails at least once a week
* Adults with any of the following diagnoses: asthma, allergic rhinitis, atopic eczema, migraine, tension headache, depression
* Adolescents with any of the following diagnoses: asthma, allergic rhinitis, atopic eczema
* informed written consent

Exclusion criteria:

* Participation in a disease-management program
* Participation in an intervention study
* Cancer diagnosis
* current usage of a complementary therapy (control group only)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Insured people of the statutory health insurance Techniker Krankenkasse in Germany
Sampling Method: Non-Probability Sample
Enrollment: 3960 (Actual)
Dates: Start 2013-03; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis-specific patient reported outcomes | 6 months
  Questionnaires:
  asthma: AQLQ, (PAQLQ for adolescents) allergic rhinitis: RQLQ (AdolRQLQ for adolescents) atopic eczema: DLQI (CDLQI for adolescents) migraine and headache: days with headache (last 4 weeks) tension headache: days of headache within the last 4 weeks

SECONDARY OUTCOMES:
Health related quality of life (SF-12) | 3, 6 and 12 months
Costs | 3, 6, and 12 months period
Diagnoses-specific patient reported outcomes | 3 and 12 months
  same parameters as for primary outcome, but different time point

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, MBA, Principal Investigator — Charite Universitätsmedizin Berlin; Thomas Reinhold, PhD, Principal Investigator — Charite-Universitätsmedizin Berlin
Locations (1):
- Institute for Social Medicine, Epidemiology and Health Economics Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Kass B, Icke K, Witt CM, Reinhold T. Effectiveness and cost-effectiveness of treatment with additional enrollment to a homeopathic integrated care contract in Germany. BMC Health Serv Res. 2020 Sep 15;20(1):872. doi: 10.1186/s12913-020-05706-4. PMID 32933511